CLINICAL TRIAL: NCT01306656
Title: Randomized Controlled Trial of Vitamin D Repletion Regimens in Primary Hyperparathyroidism
Brief Title: Vitamin D Repletion in Primary Hyperparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shonni J. Silverberg, Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAF1797; R01DK084986-05 (NIH)
Record Dates: First submitted 2011-02-10; First posted 2011-03-02 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Primary Hyperparathyroidism; Vitamin D Deficiency
Keywords: Endocrinology; Metabolic Bone Disease; Primary Hyperparathyroidism; PHPT; Vitamin D Deficiency; Bone Mineral Density; Hyper-calcemia
MeSH Terms: conditions — Hyperparathyroidism, Primary; Vitamin D Deficiency; Bone Diseases, Metabolic | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: Active arm:
  Month 1: 20,000 IU vitamin D3 once a week, plus daily multivitamin with 400 IU vitamin D.
  Months 2-6: 10,000 IU vitamin D3 once a week, plus daily multivitamin with 400 IU vitamin D.
  Placebo arm:
  Month 1: Placebo once a week plus daily multivitamin with 400 IU vitamin D.
  Months 2-6: Placebo every week plus daily multivitamin with 400 IU vitamin D.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patient, investigator and study team will be blinded to study arm ramdomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): 10,000 IU Vitamin D3 plus a multivitamin with 400 IU vitamin D
  Interventions: Drug: 10,000 IU Vitamin D3; Dietary Supplement: Vitamin D
- Group 2 (Placebo Comparator): Placebo plus a multivitamin with 400 IU vitamin D
  Interventions: Other: Placebo; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: 10,000 IU Vitamin D3 — Month 1: 20,000 IU vitamin D3 once a week
  Months 2-6: 10,000 IU vitamin D3 once a week
  Other Names: Cholecalciferol-D3
  Arms: Group 1
Other: Placebo — Month 1: Placebo once a week
  Months 2-6: Placebo once a week
  Other Names: Placebo pill
  Arms: Group 2
Dietary Supplement: Vitamin D — Daily multivitamin with 400 IU vitamin D.
  Other Names: cholecalciferol

SUMMARY:
This study will look at the effect of 2 treatment regimens that contain vitamin D in a six-month treatment trial of patients with PHPT who are vitamin D deficient. Patients will be assigned randomly to one of 2 regimens, and will be followed with tests of their blood, urine and bones. This study should provide important information on the effect of vitamin D therapy in patients with PHPT. In addition, data from this study will guide physicians as to how best to treat their patients who have PHPT and vitamin D deficiency.

DETAILED DESCRIPTION:
Primary hyperparathyroidism (PHPT) is a common disease in which the parathyroid glands produce excessive amounts of parathyroid hormone (PTH), which regulates calcium levels. In primary hyperparathyroidism, high levels of PTH remove too much calcium from bones and deposit the excess calcium in the blood, which is then filtered into the urine by the kidneys. Bone health is threatened by the excess calcium loss which weakens the structure of the bones.

Many patients with primary hyperparathyroidism also have low vitamin D (25OHD) levels which is thought to further impair bone health. Recent medical guidelines recommend treating patients with primary hyperparathyroidism who have low vitamin D levels with oral vitamin D but the optimal vitamin D dose and rate of repletion is unclear. It is, therefore, important to determine if replenishing Vitamin D will improve bone health in primary hyperparathyroidism, and if so, to assess the impact of the rate of vitamin D repletion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PHPT, defined by an elevated serum calcium level (we will not study normocalcemic PHPT) with elevated or inappropriately normal PTH levels.
* Vitamin D3 less than 30 ng/ml

Exclusion Criteria:

* Patients with familial hyperparathyroid syndromes
* Current or past use of the following medications: bisphosphonate within past 2 years, use of lithium or thiazide diuretics, current use of cinacalcet, use of aluminum containing medications, cimetidine, colestipol, or orlistat
* Malignancy, except cured basal or squamous cell skin carcinoma or other cured cancers that are at least five years free from recurrence
* History or current diagnosis of certain medical diseases (including sarcoidosis, active infectious granulomatous disease, HIV/AIDS, chronic kidney disease (serum creatinine > 1.5 mg/dL), liver disease; GI diseases known to affect calcium metabolism; secondary hyperparathyroidism);
* We will also exclude patients with calcium above 11.5 mg/dL, urine calcium above 350 mg/day, and active nephrolithiasis because vitamin D repletion could potentially exacerbate hypercalcemia or hypercalciuria
* Other exclusions include protected individuals (institutionalized), prisoners, and any other prospective participant who might not be able to give voluntary informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shonni J Silverberg, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 10,000 IU Vitamin D3 + Multivitamin: 10,000 IU Vitamin D3 plus a multivitamin with 400 IU vitamin D
  10,000 IU Vitamin D3: Month 1: 20,000 IU vitamin D3 once a week
  Months 2-6: 10,000 IU vitamin D3 once a week
  Vitamin D: Daily multivitamin with 400 IU vitamin D.
- Placebo + Multivitamin: Placebo plus a multivitamin with 400 IU vitamin D
  Placebo: Month 1: Placebo once a week
  Months 2-6: Placebo once a week
  Vitamin D: Daily multivitamin with 400 IU vitamin D.
Period: Overall Study
Arm/Group | 10,000 IU Vitamin D3 + Multivitamin | Placebo + Multivitamin
Started | 7 | 2
Completed | 6 | 2
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10,000 IU Vitamin D3 + Multivitamin | Placebo + Multivitamin | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Serum Parathyroid Hormone (PTH) Level
Description: This is designed to measure how many participants will achieve PTH > 65 pg/mL.
Time Frame: 6 months
Population: Study enrollment did not reach the required number of subjects; the analysis results would not have been reliable or have enough statistical power. Therefore, samples were not processed and data was not available for analysis.
Arm/Group | 10,000 IU Vitamin D3 + Multivitamin | Placebo + Multivitamin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Areal Bone Mineral Density of the Lumbar Spine
Description: Measured by dual-energy x-ray absorptiometry (DEXA) scan
Time Frame: 6 months
Population: Study enrollment did not reach the required number of subjects; the analysis results are not reliable or have enough statistical power.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | 10,000 IU Vitamin D3 + Multivitamin | Placebo + Multivitamin
Number analyzed (Participants) | 6 | 2
percentage of change | -.98777 (1.662643) | 1.442861 (4.376592)

3. Secondary Outcome: Trabecular Bone Density at the Forearm
Description: Measured by high resolution peripheral quantitative computed tomography
Time Frame: 6 months
Population: Study enrollment did not reach the required number of subjects; the analysis results are not reliable nor have enough statistical power.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Group 1: 10,000 IU Vitamin D3 plus a multivitamin with 400 IU vitamin D
  10,000 IU Vitamin D3: Month 1: 20,000 IU vitamin D3 once a week
  Months 2-6: 10,000 IU vitamin D3 once a week
  Vitamin D: Daily multivitamin with 400 IU vitamin D.
- Group 2: Placebo plus a multivitamin with 400 IU vitamin D
  Placebo: Month 1: Placebo once a week
  Months 2-6: Placebo once a week
  Vitamin D: Daily multivitamin with 400 IU vitamin D.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 2
percentage of change | -1.00345 (3.912386) | -2.59816 (0.583978)

4. Secondary Outcome: Change in Urinary Calcium Level
Description: This is designed to measure how the study treatment will affect urinary calcium level over time.
Time Frame: 1 month, 3 months, 6 months
Population: Data is provided for 6 out of the 7 participants in Group 1 due to that 1 participant became lost to follow-up and did not complete lab testing at Month 3 and 6.
Measure: Mean (Full Range); unit: mg/day
Arm/Group | 10,000 IU Vitamin D3 + Multivitamin | Placebo + Multivitamin
Number analyzed (Participants) | 6 | 2
mg/day
  1-month | 182.67 [9 to 453] | 154 [76 to 232]
  3-month | 172.67 [6 to 282] | 115.5 [51 to 180]
  6-month | 195.17 [12 to 387] | 50.5 [30 to 71]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definitions do not differ from those of the ClinicalTrials.gov definitions.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 1/7 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=7) | Group 2 (N=2)
Infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary infection - E. Coli
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Constipation for 5 days
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0) — right nephrolithiasis

LIMITATIONS AND CAVEATS:
Study enrollment did not reach the required number of subjects; the analysis results would not have been reliable or have enough statistical power. Therefore, samples were not processed and data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT01306656/Prot_SAP_000.pdf